CLINICAL TRIAL: NCT02789241
Title: Dose-Related Inflammatory Effects of Intravenous Endotoxin in Humans: An Evaluation of a New Clinical Lot of Escherichia Coli (E. Coli Group O 113:H10:K Negative) Endotoxin in Healthy Volunteers
Brief Title: Dose-Related Inflammatory Effects of Intravenous Endotoxin in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert J Noveck, M.D. (Other)
Collaborators: Foundation for the National Institutes of Health (Other)
Responsible Party: Sponsor-Investigator, Robert J Noveck, M.D., Associate Professior and Co-Director, Division of Clinical Pharmacology and Medical Director, Duke Clinical Research Unit, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00070829
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Endotoxin; healthy; volunteers; males; females
MeSH Terms: interventions — Endotoxins; Lipopolysaccharides; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endotoxin (LPS) (Experimental): The safety and tolerability will be assessed at different doses that will consist of 4 groups; each consisting of 4 subjects receiving endotoxin (LPS). Group 1 will test the low dose of LPS (0.6 ng/kg); Group 2 will test the 1.0 ng/kg dose; Group 3 will test the 2.0 ng/kg dose and Group 4 will test the 4.0 ng/kg dose.
  Interventions: Biological: Endotoxin
- Placebo (Placebo Comparator): The trial will consist of 4 groups each group will have 2 subjects receiving Placebo (normal saline)].
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Endotoxin — Reference Endotoxin is a purified LPS prepared from Escherichia coli O:113 (US Standard Reference Endotoxin); Clinical Center Reference Endotoxin (CCRE) Lot #94332B1 manufactured and vialed under GMP guidelines by List Biological Labs, Inc., 540 Division St., Campbell, CA 95008, for the Pharmacy Development Service, Clinical Center, National Institutes of Health, Bethesda, MD, USA. The material has been approved by the FDA (Food and Drug Administration) for 'Investigational Use Only'. This specific Lot from List Biological Labs specified for use in this study contains 1 mcg/vial.
  Other Names: LPS; Lipopolysaccharide; Reference Endotoxin; CCRE; CCRE Lot 94332B1
  Arms: Endotoxin (LPS)
Other: Placebo — Normal saline will be administered as the control to evaluate the effects on the biomarkers over time and to compare the responses following LPS to those following the control injection of normal saline.
  Other Names: Normal Saline (NS); Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate 4-dose levels of CCRE Lot 94332B1 (0.6, 1.0, 2.0, and 4.0 ng/kg). This study is known as, an "endotoxin challenge." Thousands of healthy subjects worldwide over the last 20 years have participated in endotoxin challenge studies as part of clinical research and clinical drug development programs. This study will only test the safety and tolerability of CCRE Lot 94332B1.

DETAILED DESCRIPTION:
Normal healthy subjects will be recruited and consented for the study. Following completion of the study, the bio-marker samples will be sent to Dr. Anthony Suffredini a collaborator and Deputy Chief & Senior Investigator Department of Critical Care Medicine at the National Institutes of Health (NIH). All samples will be de-identified and analyzed at the NIH; the results of which will be reviewed by both Drs. Suffredini and Noveck. Statistical analysis will be performed at the NIH by the Department of Statistics from which manuscripts will be written for publication.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between the ages of 18-40 years, inclusive, at the time of Informed Consent. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Agreement by female subjects with reproductive potential to be using an adequate method of contraception and agrees to continue using this method for the duration of the study. Female subjects must also agree to the use of TWO reliable methods of contraception following receiving study drug; if sexually active, which can include: condoms, spermicidal gel, diaphragm, hormonal or non-hormonal intrauterine device, surgical sterilization, an oral contraceptive pill (OCP), and depot progesterone injections.
* Body Mass Index (BMI) of 18-32 kg/m2 and a total body weight >50 kg (110 lb), but <95 kg.
* The subject has demonstrably adequate veins for IV catheter insertion.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all the pertinent aspects of the study.
* Subjects who are willing and able to comply with the scheduled visits, laboratory tests, and other study procedures.
* Male subjects agree that they [or their female partner(s)] will use an acceptable contraceptive regimen throughout the duration of the study. Acceptable contraception for a subject (or female partner) is being surgically sterilized; or willing to use condoms plus contraceptive foam or jelly (with all female partners who are not surgically sterilized).
* The subject has the ability and willingness to comply with protocol requirements during the study, including fasting and refraining from alcohol, nicotine and caffeine consumption from 48h prior to check-in until discharge from the unit.
* On the morning of endotoxin, Study Day 1, prior to dosing, the subject must have a normal stable baseline body temperature defined as the average of three consecutive oral temperatures (recorded, repeatedly, approximately every 10-15 seconds) between 97.0 degrees F (36.1°C) and 98.8 degrees F (37.1°C) and do not differ by >0.4 degrees F (>0.2 degrees C).
* The subject has a high probability for compliance with and completion of the study.

Exclusion Criteria:

* Evidence or history of clinically significant dental (presence of abscess), hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* A positive urine drug test for cannabinoids, amphetamines, barbiturates, cocaine, opiates, benzodiazepines, phencyclidine, and/or methadone and alcohol (breathalyzer) test at either Screening or Day -1.
* History or evidence of habitual use of tobacco- or nicotine-containing products within 3 months of screening.
* A positive serum pregnancy test (females only) at Screening or a positive urine pregnancy test at check-in.
* Subjects who have previously received endotoxin (LPS) within the previous 6 months or known hypersensitivity to endotoxin at any time.
* Subjects who have experienced cold/flu symptoms (i.e., runny nose, cough, and/or fever) or received any antibiotic treatment within 30 days or has undergone a surgical procedure within 60 days prior of the endotoxin challenge
* History of recurrent or chronic infections of any type such as tuberculosis, sinusitis, urinary tract infection, respiratory tract or dental (abscess) infection, etc. Also excluded are subjects with recurrent oral or genital herpes, recurrent herpes zoster, or any infection otherwise judged by the investigator to have the potential for exacerbation by participation in the study.
* History of syncope or symptoms of lightheadedness associated with blood draws
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening or history of drug use within 12 months prior to study drug administration, which the Investigator considers abusive.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives, whichever is longer, preceding the first dose of study medication. Also, if received an immunosuppressive drug or had received a vaccination within 3 months of Day 1
* Screening supine BP >140 or <100 mm Hg (systolic), or >90 or <60 mmHg (diastolic); following at least 5 minutes of rest. If BP is >140 or <100 mm Hg (systolic), or >90 or <60 mm Hg (diastolic), the BP should be repeated two more times and the median of the three systolic and the median of the three diastolic BP values should be used to determine the subject's eligibility. If either of the median values is outside of the criteria above, the subject is excluded.
* Resting heart rate (HR) at screening or check-in on Day -1 <50 bpm (beats per minute) following at least 10 minutes of rest from either vital signs or ECGs. If HR is <50 bpm, the HR should be repeated two more times and the median of the three HR values should be used to determine the subject's eligibility. If the median value is <50 bpm, the subject is excluded.
* 12 lead ECG demonstrating HR < 50 bpm, QTc >450 or a QRS interval >120 msec at screening of check-in. If the heart rate or QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the median of the three QTc values should be used to determine the subject's eligibility. If the median value for any of these parameters is outside the limit specified, the subject is excluded.
* Use of prescription or nonprescription drugs and dietary supplements, especially those with anti-inflammatory properties (e.g. fish oil, turmeric, etc.) within 7 days or 5 half-lives (whichever is longer) prior to receiving endotoxin. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis. Use of any steroidal or non-steroidal anti-inflammatory drug (NSAID) within 7 days or 5 half-lives (whichever is longer) of admission of each period is specifically prohibited due to potential confounding effects on the study PD endpoints
* History of frequent headaches (>2 per month) or migraines or headaches from an absence of caffeine from coffee, tea, chocolate, or other caffeine-related substances
* Caffeine consumption in excess of 3 cups per day
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* Women who are of non-childbearing potential must be:

  1. Surgically sterile (removal of both ovaries and/ or uterus at least 12 months prior to dosing).
  2. Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing on Day -1 and with an FSH level at screening of ≥ 40 mIU/mL.
  3. Women of child-bearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy at check-in, and must agree to avoid pregnancy during study. Pregnancy is tested at screening, during check-in, and at any given time if deemed necessary by the PI or designate. During the study, women of child-bearing potential must use two acceptable methods of contraception at the same time. Medically acceptable contraceptives include: (1) documented surgical sterilization (such as a hysterectomy), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or the use of a condom with a spermicide and (3) hormonal contraception (combination oral contraceptives, transdermal patch, injectables, implantables or vaginal ring) or (4) an intrauterine device (IUD) or intrauterine system (IUS). Abstinence is not an acceptable form of contraception in this study.
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator directly involved in the conduct of the study.
* The subject has a clinically significant abnormal white blood cell (WBC) count, differential or presence of clinically significant WBCs on the microscopic examination of the urinalysis.
* The subject has engaged in sunbathing or in any physical exercise, sports or exertion other than normal walking within 72h of check-in
* The subject has an elevated temperature, presence of dental/other abscess, chills, malaise, cough, cold, and/or headache which are suggestive of an occult infection (viral, bacterial, etc.).
* The subject has donated more than 250 mL of blood within 30 days of Day 1 or has donated more than 500 mL of blood within 56 days of Day 1
* The subject has a known allergy/sensitivity to lactose and/ or polyethylene glycol (excipients in the LPS injection).
* Pregnant or breastfeeding females.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in heart rate | Baseline, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5, 5.75, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, and 24 hours after the LPS administration
  Safety will be assessed by measuring heart rate.
Number of treatment emergent adverse events (TEAEs) | every 15 minutes for up to 6 hours
Change in blood pressure | Baseline, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5, 5.75, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, and 24 hours after the LPS administration
  Safety will be assessed by measuring blood pressure
Change in ECG parameters | Baseline, 1, 2, 4, 8, and 24 hours after LPS administration
Change in respiratory rate | Baseline, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5, 5.75, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, and 24 hours after the LPS administration
  Safety will be assessed by measuring respiratory rate
Change in body temperature | Baseline, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5, 5.75, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, and 24 hours after the LPS administration
  Safety will be assessed by measuring body temperature
Change in Pulse Oximetry | Baseline, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5, 5.75, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, and 24 hours after the LPS administration
  Safety will be assessed by measuring pulse oximetry
Dose-Response Comparison | Baseline, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after LPS administration.
  Comparisons between the LPS doses and their responses will be assessed

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) | Baseline, 2-6, and 24 hours after LPS administration.
Change in Affect Rating Scale | Baseline, 2-6, and 24 hours after LPS administration.
Change in plasma pro-inflammatory cytokines | Baseline, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after LPS administration.
Change in RNA | Baseline, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after LPS administration.
Change in hsC-reactive protein | Baseline, and at approximately 24 hours after LPS administration.
Change in cortisol levels | Baseline, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after LPS administration.
Change in complete blood count | Baseline, 1, 2, 4, 6, 8, 12 and 24 hours after LPS administration.
Change in WBC counts | Baseline, 1, 2, 4, 6, 8, 12 and 24 hours after LPS administration.
Change in lymphocytes | Baseline, 1, 2, 4, 6, 8, 12 and 24 hours after LPS administration.
Change in monocytes | Baseline, 1, 2, 4, 6, 8, 12 and 24 hours after LPS administration.
Change in mRNA | Baseline, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after LPS administration.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Noveck, MD, PhD, Principal Investigator — Medical Director, Duke Early Phase Clinical Research (DEPRU)
Locations (1):
- Duke Early Phase Clinical Research (DEPRU), Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The bio-marker specimens collected will be shipped to the NIH for analysis and reviewed by the investigator and Dr. Anthony Suffredini who is a collaborator on the trial and is the Deputy Chief & Senior Investigator in the Department of Critical Care Medicine at the National Institutes of Health